CLINICAL TRIAL: NCT05573087
Title: Comparing Land-based and Aquatic Reduced Exertion High Intensity Interval Training in Sedentary Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Miriam Leary, PhD RCEP, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1911776700
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Physical Performance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquatic Based Exercise (Active Comparator): maximal jump squats in a pool
  Interventions: Other: Aquatic Based Exercise
- Land Based Exercise (Active Comparator): cycle ergometer
  Interventions: Other: Land Based Exercise

INTERVENTIONS:
Other: Aquatic Based Exercise — 10 minutes of exercise with two 20 second sprints three days per week for 8 consecutive weeks
  Arms: Aquatic Based Exercise
Other: Land Based Exercise — 10 minutes of exercise with two 20 second sprints three days per week for 8 consecutive weeks
  Arms: Land Based Exercise

SUMMARY:
Previous research has found improvements in performance (VO2max) and clinical (insulin resistance) with cycling REHIIT. In some populations (e.g. obese, arthritic) aquatic exercise is a safer, more enjoyable option. However, to date, no study has yet examined whether aquatic REHIIT confers the same benefits as land-based REHIIT. Therefore, the purpose of this study is to determine whether there are significant differences in clinical and performance outcomes between a land-based and comparable aquatics based Reduced Exertion High Intensity Interval Training (REHIIT) protocol.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* sedentary individuals; Sedentary will be defined as less than 150 minutes of exercise/week as defined by the CDC and American College of Sports Medicine
* All subjects will be screened with a resting 12 lead EKG to ensure they are safe to exercise

Exclusion Criteria:

* Any vulnerable populations will be excluded including adults unable to consent/Cognitively Impaired
* individuals who are not yet adults
* pregnant or nursing women
* prisoners or other detained individuals

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in Cardiorespiratory Fitness | Baseline to 8 weeks
  Percent changes in VO2 is milliliters of oxygen per kilogram of body weight per minute (oxygen in milliliters, weight in kilograms, and time in minutes and expressed in ml/kg/min).

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Leary, PhD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States